CLINICAL TRIAL: NCT06572969
Title: Effect of 8-week Incremental Elastic-Resistance Kick Training in Taekwondo Athlete's: Roundhouse Kick Quality and Physical Performance Analysis
Brief Title: Effect of 8-week Incremental Elastic-Resistance Kick Training in Taekwondo Athlete's
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bruno Figueira (Other)
Responsible Party: Sponsor-Investigator, Bruno Figueira, Principal Investigator, University of Évora
Organization: University of Évora (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: #SA-EK-23-29
Record Dates: First submitted 2024-08-20; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Strength; Performance
Keywords: Youth; Performance; Strength

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): In the experimental group, participants performed the RHK exercises using incrementally resistive elastic tubing. The RHKs targeted shields (Adidas, Curved Kick Shield) held at chest height. Each athlete started with a 2.4 m elastic tubing, one end attached to the ankle and the other to a stable platform, ensuring the tubing's resistance reached 50 N at full kicked extension (Fig.1). After four weeks (12 sessions), resistance increased to 100 N by adding another tubing. Each session comprised three sets of 6 RHKs per leg, at maximum speed, with 30-second intervals between kicks and 3-minute rests between sets. This 8-week, three times weekly, training regimen involved incremental ER training.
  Interventions: Other: Elastic-Resistance Kick Training
- Control (Other): The control group undertook a similar RHK training regime in sequence and duration, mirroring the number of kicks performed by the experimental group, but without ER equipment. After each training session, a 5-minute rest allotted before resuming standard Taekwondo training. Post the 8-week training, both groups underwent a 2-week retention period with uniform training program.
  Interventions: Other: No Elastic-Resistance Kick Training

INTERVENTIONS:
Other: Elastic-Resistance Kick Training — Athletes used tailored Elastic Resistance training
  Arms: Experimental
Other: No Elastic-Resistance Kick Training — Regular Taekwondo regimen without Elastic Resistance training
  Arms: Control

SUMMARY:
This study aimed to assess the effects of an 8-week incremental elastic-resistance kick training program on the roundhouse kick quality and physical performance, in comparison to conventional training methods of youth Taekwondo athletes. A two-group parallel, randomized, quasi-experimental design was used, dividing Participants into experimental (n=11, age: 15.5 ± 1.5 years, stature: 169.5 ± 15.5 cm, body mass: 63.2 ± 26.2 kg; training experience: 7.0 ± 3.0 y) and control group (n=10, age: 14.8 ± 1.2 years, stature: 162.0 ± 14.0 cm, body mass: 53.15 ± 21.4 kg; training experience: 5.5 ± 1.5 y), undergoing tailored Elastic Resistance training alongside their regular Taekwondo regimen. The study measured various performance metrics including Roundhouse Kick velocity, impact scoring, isometric muscle strength, counter movement jump performance, and simple reaction times.

ELIGIBILITY:
Inclusion Criteria:

* Being part of a unified youth development program;
* Minimum of four weekly training sessions, each session lasting 90 minutes.

Exclusion Criteria:

* Musculoskeletal, neurological, or orthopedic injury that may impair their participation.

Ages: 14 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 37 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-03-10 (Actual); Study Completion 2024-03-20 (Actual)

PRIMARY OUTCOMES:
kick velocity | 8 weeks
  subjects executed three maximal RHKs with each leg, taking a 20-second rest between kicks. The best performance time was recorded.

SECONDARY OUTCOMES:
Simple Eye-Hand Reaction Time Test | 8 weeks
  For E-H reaction measurements, participants sit about 50 cm from the computer screen, with the screen placed 15 cm in front of and at the same height as the response panel. The response involves using the index finger of one hand, with the other hand resting beside the panel.

OTHER OUTCOMES:
Eye-Foot Reaction Time Test | 8 weeks
  Simple Eye-foot (E-F) reactions were measured similarly, with the participant seated the same distance from the screen. The response panel is placed on the floor, positioned under the seated subject's foot. The response is made using the toe, while both hands rest on the desk and the other leg is positioned next to the panel.
Back-Leg-Chest Muscle Strength Dynamometry | 8 weeks
  Participants, free from lifting restrictions, underwent Isometric Muscle Strength (IMS) testing using a back-leg-chest dynamometer (Saehan, SH5007, Masan 630-728, Korea). This device, correlated (r = 0.77, p <.001) with manual muscle tests 29, measures force applied to a spring, moving a pointer to indicate the exerted force. The dynamometer records up to 300 kg with 1 kg resolution, accurate to + 0.5 kg at 100kg. Subjects were instructed to stand with a 30-degree knee flexion and hip flexion, maintaining a proper lordotic curve, and then exert force using their legs and arms. The average of two strength measurements at each testing phase distinguished between learning and training effects. Participants controlled the exertion level, with to avoid discomfort.
Margaria-Kalamen Anaerobic Alactic Power Test | 8 weeks
  The Margaria-Kalamen stair climb test measures an athlete's lower body peak power 30. Participants start 5 meters away from the first stair, quickly ascending on the researcher's signal, taking three steps at a time. Timers on the 3rd and 9th steps record the duration of the climb, starting and stopping as the participant hits these steps. The best performance time from three trials, each followed by a 20-second rest, is used. Anaerobic power, calculated in watts, is derived by multiplying the participant's weight by the stair height (16 steps) and gravitational acceleration (9.81 m·sec-1), and dividing by the time taken. This formula for computing anaerobic-alactic power follows 31:
  Equation: Anaerobic Alactic Power (watts) = (body mass (kg) × distance (0.96 m) × 9.81m·sec-1) / time (sec-1).
10 m Sprint test | 8 weeks
  In the 10 m sprint test (S-10m), participants completed three maximum-effort 10-meter sprints, timed using a Brower equipment (Wireless Sprint System, Draper, UT, USA). Photocells were placed at the start line (0 m) and at the 10 m mark, positioned 1 meter above the floor, aligning with the manufacturer's standard tripod height. Sprints were interspersed with 3-minute rest periods, and the fast sprint was recorded. This system validity and reliability have been confirmed, demonstrating an intraclass correlation coefficient between 0.92 and 0.98 and a coefficient of variation of 1.6% 32.
Jump Performance Test | 8 weeks
  Lower limb power was evaluated using the counter movement jump (CMJ) test. Participants began each CMJ from a static standing position, executing a countermovement and then a rapid extension of the lower limb. They perform three maximal effort CMJ's, with 90-second rest intervals between jumps. The countermovement phase was self-selected, allowing athletes to use their preferred jumping technique. Participants were instructed to keep their trunk vertical and hands on their hips during jumps. Data was captured using an iPhone 11 Pro with My Jump app 27, recording at 240 frames per second.

CONTACTS AND LOCATIONS:
Locations (1):
- Bruno Figueira, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP